CLINICAL TRIAL: NCT05168397
Title: Evaluation of the Cutaneous and Ocular Tolerance of RV4857A Sunscreen Product and Its Efficacy Against the Recurrence of Lesions Post Sun Exposure in Subjects With Facial Acne
Brief Title: Sunscreen Efficacy Against the Reccurence of Lesions Post-sun Exposure in Acneic Subjects
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV4857A202092
Record Dates: First submitted 2021-09-29; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Acne
Keywords: Sunscreen; Lesions post sun exposure; Anti-imperfections
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RV4857A arm: Application of the product before and during each sun exposure, at least twice a day.
  During sun exposures, the applications were renewed as often as necessary, in particular after swimming, perspiring, towelling, in order to ensure a good protection. On days of bad weather, the product was applied in the morning and at the beginning of the afternoon.
  Interventions: Other: RV4857A

INTERVENTIONS:
Other: RV4857A — RV4857A formula CD2110 is a sunscreen product

SUMMARY:
The aim of this study is firstly to assess the tolerance of the sunscreen RV4857A-CD2110 after 28 days and 57 days of at least a twice daily on the study areas, secondly to assess anti-imperfection efficacy after 28 days and 57 days of use and its efficacy against recurrence of acne lesions post-sun exposure.

DETAILED DESCRIPTION:
This is a monocentric study on adults and adolescents with acne prone skin on the face. This open-labelled study aim first to assess the dermatological and ophthalmological tolerance of the investigational sunscreen product RV4857A formula CD2110 after 28 days and, dermatological tolerance after 57 days of at least a twice daily on the study areas, under normal conditions of use, on 40 subjects intending to have a minimum of 10 days per month of sun exposure duration ≥ 1h, in the time slot 11am-4pm and intending to have a minimum of 4 swimming sessions (sea or swimming pool) during at least the first month of the study.

Secondary objectives :

* To assess the anti-imperfection efficacy of the product during the summer
* To assess the "non" rebound effect (non recurrence of acne) one month after stopping the application of the sunscreen and without any sun exposure at D85 (difference between D85 and D0)
* To evaluate the impact on Quality of Life of subjects through CADI and DLQI questionnaires (or CDLQI questionnaire for adolescent from 12 to 16 years-old) completed at baseline, D29 and D57

The study includes 4 visits :

* Visit 1: Inclusion visit (D1)
* Visit 2: Intermediate visit (D29)
* Visit 3: Intermediate visit "end of summer" (D57), a Stop the application of the sunscreen product (and stop sun exposure) between Visit 3 and the end of the study Visit 4: End of study visit in autumn (D85)

The theoretical study duration for each subject will be 85 days with at least 57 days of product use. The study interest areas are Face and Neck.

ELIGIBILITY:
Inclusion Criteria:

1. Related to the population:

   * Females and/or males (with at least 25% of male)
   * Age: adults from 18 to 40 years old and adolescent from 12 to 17 years old (33% to 50% of the total population)
   * Considered "healthy subject" by the Investigator
   * Being of Phototype I to IV
   * Subject with combination to oily skin
   * Subject who foresees sun exposure during the first 2 months of the study
   * Subjects must be registered with health social security or health social insurance (if required by national regulations)
   * Subject and/or parent(s)/legal representative(s) who have signed his/her/their written informed consent for his/her participation in the study (or his/her/their child participation in the study) and a photograph authorization
   * For woman of childbearing potential: committing herself to use effective contraceptive method since at least 3 months before the beginning of the study and committing to it throughout the study
   * Regular users of very high protection sunscreen products.
2. Related to the disease:

   * For adults and adolescents: subject with mild to moderate acne with a total of 10 to 40 acne lesions (at least 5 non-inflammatory lesions (open and closed comedones) and at least 3 to 10 inflammatory lesions (papules and pustules) maximum on the face, excluding the nose area), at the inclusion.
   * Subject prone to have recurrence of acne lesions in autumn (declarative)

Exclusion Criteria:

1. Related to the population:

   * Having participated in another clinical trial within 4 weeks before the inclusion visit and for a longer period if required in the Investigator's opinion Taking part or planning to participate in another clinical trial during the study in the same or another investigation centre
   * Breastfeeding or pregnant or not willing to take necessary precautions to avoid pregnancy during the study and for at least 3 months before the inclusion visit (for the woman of childbearing potential)
   * Subject or parent(s)/legal representative(s) deprived of freedom by administrative or legal decision or under guardianship
   * Subject or parent(s)/legal representative(s) not able to be contacted in case of emergency
   * Subject admitted in a sanitary or social facility
   * Subject planning a hospitalization during the study
2. Related to the disease

   * Cutaneous pathology (psoriasis, atopic dermatitis, skin infectious disease of viral, bacterial, fungus or parasitic origin …) or dermatological condition (especially pityriasis versicolor, severe pigmentation disorders) on the studied zone other than acne liable to interfere with the data of the study
   * Severe acne
   * Clinical signs of hormonal disfunctions or hyperandrogenism
   * Excessive exposure to sunlight or UV-rays within the previous month
   * Having history of abnormal reactions from exposure to sunlight
   * Use of self tanning product during the previous month History of hypersensitivity or intolerance to any cosmetic product
3. Related to treatments

   * Use of a systemic or topical medication with anti-inflammatory or photosensitising products during the previous 2 weeks and for systemic medication with corticoids and/or antihistaminics during the previous 4 weeks
   * Use of a systemic treatment for acne during the previous month for antibiotics, zinc gluconate and hormonal treatment and during the 6 previous months for isotretinoin
   * Use of a topical treatment for acne during the previous month (benzoil peroxide, retinoid, antibiotics, azelaic acid…)
   * Use of anti-acneic or anti-seborrheic cosmestic care (containing alpha hydroxy-acids, retinoic derivatives..) during the 15 previous days
   * Use of other topical or systemic treatment during the previous weeks liable to interfere with the assessment of the cutaneous tolerance and efficacy of the studied product (according to the investigator's appreciation)
   * Any surgery, chemical or physical treatment on the experimental area within the 12 months prior to the study or foreseeing it for the duration of the study
   * Woman whose oral contraception is instaured or changed for less than 3 months

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be recruited from the investigation centre's panel. The participants will be selected on the basis of inclusion and non-inclusion criteria specific to the study and on their ability to comply with the constraints required by the protocol. The participants will be definitely included in the study after a specific interview and a clinical examination
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Assessment of the dermatological physical signs | Change from Baseline to 30 minutes after product application, to 29 and 57 days later
  The assessment of the dermatological physical signs is based on a visual examination
Assessment of the dermatological functional signs | Change from Baseline to 30 minutes after product application, to 29 and 57 days later
  The functional signs is assessed by questioning the subject
Assessment of the ophthalmological physical signs | Change from Baseline to 30 minutes after product application, to 29 and 57 days later
  The assessment of the ophthalmological physical signs is based on a dermatologist visual examination
Assessment of the ophthalmological functional signs | Change from Baseline to 30 minutes after product application, to 29 and 57 days later
  The functional signs is assessed by questioning the subject
Assessment of the Tear film Break Up Time (BUT) | Change from Baseline to 30 minutes after product application, to 29 and 57 days later
  The tear film break-up time is a test to measure the relative stability of the pre-corneal tear film. This examination is performed by the same Ophthalmologist thanks to a biomicroscope after blinking (using a chronometer). The measured time will be expressed in seconds
Assessment of global tolerance assessment (dermatogical assesment), a 5-point scale | Change from Baseline to 29 and 57 days later
  * Excellent: no functional nor physical signs related to the investigational product observed or reported by the subjects
  * Very good
  * Good
  * Moderate
  * Bad
Assessment of global tolerance assessment (ophthalmological assessment), a 5-point scale | Change from Baseline to 29 days later
  * Excellent: no functional nor physical signs related to the investigational product observed or reported by the subjects
  * Very good
  * Good
  * Moderate
  * Bad

SECONDARY OUTCOMES:
Change of the number of total acne lesions on the face | Change from Baseline to 29, 57 and 85 days later
  by counting according to the method of Lucky
Change of the number of non-inflammatory lesions (open and closed comedones) on the face | Change from Baseline to 29, 57 and 85 days later
  by counting according to the method of Lucky
Change of the number of inflammatory lesions (papules, pustules, nodules) on the face | Change from Baseline to 29, 57 and 85 days later
  by counting according to the method of Lucky
Assessment of the non-comedogenic potential | Change from Baseline to 29 days later
  by statistical comparison of open and closed comedones counted by the investigator on the face before and after 28 days of application of investigational product
Change of the acne severity, assess by Global Acne Evaluation (GEA) on a 6-point scale | Change from Baseline to 29, 57 and 85 days later
  * 0: Clear
  * 1: Almost clear
  * 2: Mild
  * 3: Moderate
  * 4: Severe
  * 5 : Very Severe
Evaluation of the global acne evolution on a 6-point scale | Change from Baseline to 29 and 57 days later
  -1: Worsening, 0: No change,
  1. Mild improvement,
  2. Moderate improvement,
  3. Good improvement,
  4. Very good improvement
Evaluation of the global product efficacy by the subjects themselves regarding rebound effect in Autumn | Change from Baseline to 85 days later
  Questions Q24 and Q25 at D85 in the self-questionnaire
Assessment of the cosmetic acceptability and perceived efficacy of the product | Change from Baseline to 29 and 57 days later
  The self subject assemsment consists of different questions concerning participants' perception of the product's efficacy (majority of scales ranging from 0 to 10 where 0 was the worst satisfaction and 10 the best one)
To evaluate the impact on Quality of Life of subjects through questionnaires | Change from Baseline to 29 and 57 days later
  Quality of Life questionnaires consist of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Contreiras Pinto, PhD, Study Chair — PhD Trials®; Leonor Girão, MD, Principal Investigator — PhD Trials®
Locations (1):
- PhD Trials®, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No